CLINICAL TRIAL: NCT01201434
Title: The Effect of Probiotics on Sputum Bacteria, Sputum Inflammation, and Pulmonary Infections in Patients With Cystic Fibrosis: A Double-blind Placebo-controlled Trial
Brief Title: Effect of Probiotics on Sputum Inflammation and Pulmonary Infections in Patients With Cystic Fibrosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Severe allergic reaction in one patient
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Batia Weiss, Director, Pediatric Gastroenterology Unit, Edmond and Lily Safra Children's Hospital, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: SHEBA-10-7702-BW-CTIL
Record Dates: First submitted 2010-08-31; First posted 2010-09-14 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; probiotics; pulmonary; infections
MeSH Terms: conditions — Cystic Fibrosis; Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Probiotics, Treatment, Food Additive (Experimental)
  Interventions: Dietary Supplement: Bio-25 probiotic

INTERVENTIONS:
Dietary Supplement: Bio-25 probiotic — 2 tablets per day for 6 months
  Other Names: Bio-25 by Supherb

SUMMARY:
Patients with Cystic Fibrosis have multiple pulmonary infections and repeated antibiotic treatment. These factors taken together with high sputum viscosity and slow motility of the gastrointestinal tract-may change the pathogenicity and consistency of the intestinal pathogens. Part of the pulmonary infections in CF patients are due to intestinal pathogens. A pilot study performed by the researchers using probiotics in CF patients showed a decrease in the rate of pulmonary infections. Therefore,we planned a double-blind placebo-controlled trial to examine the effect of probiotics on pulmonary infections, sputum bacteria and sputum inflammatory markers in CF patients.

DETAILED DESCRIPTION:
Patients with Cystic Fibrosis have multiple pulmonary infections and repeated antibiotic treatment. These factors taken together with high sputum viscosity and slow motility of the gastrointestinal tract-may change the pathogenicity and consistency of the intestinal pathogens. Part of the pulmonary infections in CF patients are due to intestinal pathogens. A pilot study performed by the researchers using probiotics in CF patients showed a decrease in the rate of pulmonary infections. Therefore,we planned a double-blind placebo-controlled trial to examine the effect of probiotics on pulmonary infections, sputum bacteria and sputum inflammatory markers in CF patients. The study will be a cross-over study of probiotic and placebo arms.

ELIGIBILITY:
Inclusion Criteria:

* cystic fibrosis mild to moderate
* at least 3 pulmonary exacerbations requiring antibiotics per year
* Pseudomonas aeruginosa in the sputum
* able to produce sputum

Exclusion Criteria:

* severe pulmonary disease
* less than 3 pulmonary exacerbations per year
* unable to produce sputum

Ages: 5 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The effect of probiotics on the rate of pulmonary infections compared to placebo | October 2012
  The rate of pulmonary exacerbations requiring IV or PO antibiotic treatment during the study period in the treatment and placebo groups will be assessed.

SECONDARY OUTCOMES:
The effect of probiotics on sputum bacteria compared to placebo | October 2012
The effect of probiotics on sputum inflammatory markers | October 2012
The effect of probiotics on gastrointestinal inflammation | October 2012

CONTACTS AND LOCATIONS:
Overall Officials: Batia Weiss, MD, Principal Investigator — Pediatric Gastroenterology Unit, Edmond and Lily Safra Children's Hospital, Sheba Medical Center; Ori Efrati, MD, Principal Investigator — Pediatric Pulmonology Unit, Edmond and Lily safra Children's Hospital, Sheba Medical Center

REFERENCES:
- [Background] Weiss B, Bujanover Y, Yahav Y, Vilozni D, Fireman E, Efrati O. Probiotic supplementation affects pulmonary exacerbations in patients with cystic fibrosis: a pilot study. Pediatr Pulmonol. 2010 Jun;45(6):536-40. doi: 10.1002/ppul.21138. PMID 20503277